CLINICAL TRIAL: NCT05914974
Title: ICK-Gyn: Immunotherapy-related CRP Kinetics in Metastatic Gynecological Malignancies
Brief Title: Immunotherapy-related CRP Kinetics in Metastatic Gynecological Malignancies
Status: Recruiting | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Collaborators: University Hospital Ulm (Other); University Hospital Freiburg (Other)
Responsible Party: Sponsor
Other Study IDs: ZGynO_ICK-Gyn
Record Dates: First submitted 2023-06-13; First posted 2023-06-22 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Gynecological Malignancies; Cervical Cancer; Endometrial Cancer; Ovarian Cancer; Vulvar Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms; Ovarian Neoplasms; Vulvar Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood sample to assess laboratory parameters: Leukocytes, neutrophil granulocytes, lymphocytes, hemoglobin, hematocrit, thrombocytes, kreatinin, glomerular filtration rate (GFR), serum glutamic oxaloacetic transaminase (GOT), serum glutamic pyruvic transaminase (GPT), bilirubin, lactate dehydrogenase (LDH), thyroid stimulating hormone (TSH), fT3 (free tri-iodothyronine), fT4 (free thyroxine), amylase, CRP, biomarkers related to immune response
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group: Chemotherapy without immunotherapy
- Experimental Group: Chemotherapy in combination with immunotherapy

SUMMARY:
ICK-Gyn is a prospective, multicentric, non-interventional investigator-initiated trial (IIT) that aims to investigate the prognostic value of CRP kinetics in advanced or metastatic gynecological malignancies under immune checkpoint inhibitor (ICI) therapy on the objective response rate (ORR), progression-free survival (PFS) and overall survival (OS).

DETAILED DESCRIPTION:
Immunotherapy, which involves activating the body's immune system for cancer treatment, has already been widely incorporated into the standard care of patients with advanced and metastatic gynecological cancers.

This study aims to investigate how inflammatory markers such as C-reactive protein (CRP) change during and after immunotherapy. Study findings from other tumor types (kidney, lung, bladder) suggest that immunotherapy is particularly effective when a mild inflammatory response is triggered in the body. The investigators want to examine this using CRP measurement. CRP measurement can easily be integrated into clinical routine as it only requires a blood sample.

The goal of this prospective study is to determine whether changes in CRP levels in the blood can predict the disease progression or response to immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* women ≥ 18 years of age
* histologically proven metastatic gynecological malignancies irrespective of therapy line
* patients with advanced or metastatic gynecological malignancies must fulfill treatment requirements for ICI therapy in the experimental group
* planned ICI therapy in combination with palliative chemotherapy in the experimental group
* patients with advanced or metastatic gynecological malignancies that undergo chemotherapy without ICIs in the first therapy line in the control group
* written informed consent into ICK-Gyn

Exclusion Criteria:

* missing indication for ICI therapy in the experimental group
* any ICI therapy before inclusion into the trial
* patients with advanced or metastatic endometrial or cervical cancer in the second or higher therapy line without indication to ICI therapy
* pregnant or lactating patients
* inadequate general condition (not fit for chemotherapy)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 120 patients will be included in the study after written informed consent. Of 60 patients in the control group, which will undergo chemotherapy of physician's choice, 25 patients will be diagnosed with advanced or metastatic cervical cancer, 25 patients will be diagnosed with advanced or metastatic endometrial cancer and 10 patients will be diagnosed with advanced or metastatic ovarian or vulvar cancer.
  Of 60 patients in the experimental group, which will undergo palliative chemotherapy in combination with ICIs, 25 patients will be diagnosed with advanced or metastatic cervical cancer, 25 patients will be diagnosed with advanced or metastatic endometrial cancer and 10 patients will be diagnosed with advanced or metastatic ovarian or vulvar cancer.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2035-04 (Estimated)

PRIMARY OUTCOMES:
Prognostic value of CRP kinetics under ICI therapy on progression-free survival (PFS) | duration of therapy and follow-up data (10 years)
  Evaluation of CRP kinetics to predict progression-free survival in advanced or metastatic gynecological malignancies treated with ICIs in combination with chemotherapy. The CRP value is determined from blood samples.

SECONDARY OUTCOMES:
Prognostic value of CRP kinetics in advanced or metastatic gynecological malignancies under ICI therapy on the objective response rate (ORR) and overall survival (OS). | duration of therapy and follow-up data (10 years)
  * evaluation of CRP kinetics to predict objective response in patients with advanced or metastatic gynecological malignancies receiving ICIs in combination with chemotherapy
  * evaluation of CRP kinetics to predict overall survival in patients with advanced or metastatic gynecological malignancies receiving ICI in combination with chemotherapy
  * Exploratory analysis of further biomarkers related to immune response The respective values are determined from blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Dominik Dannehl, Dr., Principal Investigator — Department of Women's Health Tübingen
Locations (1):
- Department of Women's Health, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No